CLINICAL TRIAL: NCT06154343
Title: A Phase 1, First-In-Human, Multicenter, Open-Label,Dose-Escalation and Extension Study of GQ1005 in Subjects With HER2-Expressing Advanced Solid Tumors
Brief Title: A Study of GQ1005 in Subjects With HER2-Expressing Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GeneQuantum Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GQ1005-102
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: HER2 Expressing or Mutated Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): GQ1005 will be administered intravenously every 21 days. Dose Escalation will be guided by Bayesian Optimal Interval (BOIN) Design.
  Multiple dose grouping
  Interventions: Drug: GQ1005
- Dose Expansion (Experimental): GQ1005 at the recommended phase II dose (RP2D) will be administered intravenously every 21 days. Dose expansion will further evaluate the MTD or RP2D in different types of malignant solid tumor in four cohorts.
  Interventions: Drug: GQ1005

INTERVENTIONS:
Drug: GQ1005 — an antibody drug conjugate

SUMMARY:
This is an open-label, phase I study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of GQ1005 and preliminary anti-tumor efficacy in HER2 expressing or mutated advanced malignant solid tumor subjects.

ELIGIBILITY:
Inclusion Criteria:

The general inclusion criteria for dose escalation in Part 1 and dose expansion in Part 2 are as follows:

1. Voluntary agreement to provide written informed consent；
2. Aged 18 years or older, both male and female.
3. The expected survival time is more than 3 months.
4. ECOG performance status Score 0 or 1.
5. LVEF ≥ 50% by ECHO or MUGA scan within 28 days prior to the first dose of study drug.
6. Histologically or cytologically confirmed malignancy with at least 1 measurable lesion as assessed by RECIST v1.1.
7. Good organ function, confirmed by the following laboratory test results at Screening and within 7 days prior to the first dose of study drug:

   Platelet count ≥ 100,000/mm3; hemoglobin ≥ 9g/dL; ANC ≥ 1500/mm3; Serum CREA ≤ 1.5 × ULN, or estimated CREA clearance ≥ 60 mL/min (Cockcroft-Gault equation); ALT and AST ≤ 3 × ULN (≤ 5 x ULN if liver metastases are present); Total bilirubin ≤ 1.5 x ULN for subjects with Gilbert's syndrome or ≤ 2 x ULN for subjects with liver metastases at baseline; Prothrombin time and activated partial thromboplastin time ≤ 1.5 × ULN;
8. Adequate washout period prior to the first treatment, defined as follows:

   Major surgery ≥ 4 weeks; radiotherapy ≥ 4 weeks (≥ 2 weeks if the radiotherapy is palliative stereotactic radiotherapy without abdominal involvement); seed-radioactive therapy ≥ 3 months; Nuclein therapy ≥ 3 months; autotransplantation ≥ 3 months; Hormone therapy ≥ 2 weeks or as per investigator's judgment (breast cancer subjects) Chemotherapy or targeted therapy (including antibody drug therapy) ≥ 2 weeks (5-FU-based drugs, folinic acid preparations and/or weekly paclitaxel therapy);
   * 2 weeks (or 5 half-lives, whichever is longer) (tyrosine kinase inhibitor);
   * 4 weeks (HER2-targeted biological therapy);
   * 6 weeks (nitrosourea or mitomycin C);
   * 3 weeks (any other chemotherapy/targeted therapy);
   * 2 weeks (Chinese patent medicine with clear antitumor indication) antitumor immunotherapy ≥ 4 weeks; Any investigational drug or treatment ≥ 4 weeks; Strong inhibitors of cytochrome P450 enzyme 3A4 (CYP3A4) ≥ 1 week; Organic Anion Transport Polypeptide (OATP) Inhibitors ≥ 1 week;

   Inclusion criteria for the dose escalation phase of Part 1 only:
9. Failure of standard treatment, or intolerance, or absence of standard treatment, confirmed by pathology, HER2 expression (including IHC1+, IHC2+, IHC3+ and/or ISH*+) or subjects with advanced/unresectable or metastatic solid tumors with HER2 exon 19 or 20 mutations (non-small cell lung cancer only). If only ISH*, NGS reports are available, contact the Medical Monitor.

   Inclusion criteria for part 2a only:
10. Failure of standard treatment, intolerance, or absence of standard treatment, confirmed by pathology, HER2 overexpression (IHC 3+ or IHC 2+ and ISH* +) Advanced/unresectable or metastatic breast cancer.

    Inclusion criteria for part 2b only:
11. Advanced breast cancer with low HER2 expression, unresectable, or metastatic breast cancer that has failed standard treatment, or is not tolerated, or has no standard treatment, is confirmed by pathology. (IHC 2+ and ISH*- or ISH unknown, or IHC 1+).

    Inclusion criteria for part 2c only:
12. Non-small cell lung cancer with a HER2 exon 19 or 20 mutation that has failed, or is not tolerated, or is confirmed by a documented pathology without standard treatment.

    Inclusion criteria for part 2d only:
13. Advanced/unresectable or metastatic solid tumors with HER2 expression that have failed standard therapy, are not tolerated, or are without standard therapy, and are confirmed by pathology, with HER2 overexpression preferred. (IHC 3+ or IHC 2+ or ISH* +) Adenocarcinoma of gastric and gastroesophageal junction; Other preferred tumor types include HER2 overexpression. (IHC 3+ or IHC 2+ or ISH* +) Urothelial cancer, biliary tract cancer, endometrial cancer; Breast cancer and non-small cell lung cancer are excluded.

    * ISH+: FISH or two-color in situ hybridization (DISH).

Exclusion Criteria:

Subjects must not meet any of the following exclusion criteria to be enrolled in the study.

1. Clinically active brain metastases, defined as untreated and symptomatic, or requiring treatment with steroids or anticonvulsants to control associated symptoms. Subjects with treated asymptomatic brain metastases who do not require steroid therapy may be included in the study if they have recovered from the acute toxicity of radiation therapy.
2. Cardiovascular dysfunction or clinically significant cardiac conditions, including but not limited to:

   * Symptomatic CHF (New York Heart Association classes II to IV) or severe cardiac arrhythmia requiring treatment
   * History of myocardial infarction or troponin levels consistent with myocardial infarction (defined by the American College of Cardiology guidelines) within 6 months prior to the first dose, and unstable angina pectoris within 6 months prior to the first dose of study drug;
   * QTcF prolongation at Screening >460 milliseconds (ms) (male) and >470 ms (female) except for right bundle branch block.
3. Clinically significant acute and chronic lung disease. (e.g., interstitial pneumonia, pulmonary infection, pulmonary fibrosis, and severe radiation pneumonitis), or subjects with suspected pulmonary disease based on imaging at screening, or subjects requiring oxygen.
4. People with known hypersensitivity to recombinant humanized anti-HER2 monoclonal antibody-DXd conjugate drugs and their components or to humanized monoclonal antibody products.
5. Poorly controlled pleural, ascites, or pericardial effusions.
6. Toxicity that has not resolved from prior antineoplastic therapy, defined as toxicity (other than alopecia) that has not resolved to ≤ Grade 1 or baseline levels, is at the discretion of the investigator for the eligibility of subjects with chronic Grade 2 toxicities.
7. The prior anthracycline exposure dose met the following criteria: adriamycin > 500mg/m2; Epirubicin >900mg/m2; Pirarubicin > 950mg/m2; Mitoxanthraquinone >120mg/m2; other (i.e. liposomal doxorubicin or other anthracycline >equivalent to 500 mg/m2 of doxorubicin); If more than one anthracycline is used, the cumulative dose must not exceed the equivalent of 500 mg/m2 of doxorubicin.
8. There is an active infection requiring treatment with intravenous antibiotics, antivirals, or antifungals.
9. Known HIV infection.
10. Active hepatitis C virus infection. (HCV antibody positive and HCV-RNA higher than the upper limit of reference value); Active hepatitis B virus infection. (HBsAg positive and/or HBcAb positive and HBV-DNA quantitation ≥2000 IU/ml);, to be eligible for enrollment, subjects with chronic hepatitis B will have to agree to monthly DNA testing and receive appropriate antiviral therapy as indicated.
11. Live vaccine was administered within 30 days prior to the first dose of study drug.
12. Previous or current evidence of any concomitant disease, treatment, or laboratory abnormality that the investigator believes may confound the results of the trial or interfere with subject participation and compliance.
13. He has received treatment with an antibody-conjugated drug comprising a topoisomerase I inhibitor ezotecan derivative.
14. Breastfeeding women or women with confirmed pregnancy by a pregnancy test within 7 days prior to the first treatment.
15. Reluctant to contraception during the study and for at least 7 months after the last dose of study drug.
16. Subjects with multiple primary malignancies within the past 3 years, with the exception of fully resected non-melanoma skin cancer, cured disease in situ, cured contralateral breast cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | Up to 2 years
  Incidence and severity of Treatment-emergent adverse events, treatment-related adverse events and serious adverse events, according to NCI-CTCAE Version 5.0 (The number of participants who had treatment-related side effects in population who had received one therapy at least).
Dose Limiting Toxicities (DLTs) | From first dose to the end of Cycle 1, 21 days
  Adverse events will be assessed using NCI CTCAE version 5.0 and will be evaluated by the investigator and the sponsor for the eligibility of DLT.
Maximal Tolerance Dose (MTD) or recommended phase II dose (RP2D) | After each cohort completes the DLT observation period (Day 1 to Day 21 after the first dose of study treatment) or has a DLT or becomes not DLT-evaluable
  The SRC will also determine the MTD/RP2D based on the totality of data for all tested dose levels.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of GQ1005 | Up to2 years
  The pharmacokinetics(PK) profile of GQ1005
Time of peak plasma concentration (Tmax) | Up to2 years
  The pharmacokinetics(PK) profile of GQ1005
Area under the plasma concentration time curve (AUC) of GQ1005 | Up to 2 years
  The pharmacokinetics(PK) profile of GQ1005
Overall response rate (ORR) | Up to 2 years
  The objective response rate will be analyzed according to the RECIST 1.1 standard tumor evaluation
Duration of Response (DoR) | Up to 2 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the rate of the sum of CR, PR and SD according to the RECIST 1.1 standard tumor evaluation.
Time-to-response (TTR) | Up to 2 years
  To preliminarily evaluate TTR in patients with advanced solid tumors
Progression-free survival (PFS) | Up to 2 years
  Progression free survival (PFS) refers to the time from the date of first administration to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard
Overall Survival (OS) | Up to 2 years
  Overall survival (OS) refers to the time from the date of first administration to (for any reason) death. The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard
Immunogenicity (anti-drug antibody ADA) | Up to 2 years
  Percentage of subjects producing detectable anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Chinese PLA general hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Haerbin Medical University, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Shengjing hospital of China medical universty, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan university Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an University, Xi'an, Shangxi
  - Suining Central Hospital, Suining, Sichuan
  - Sichuan Cancer Hospital, Chengdu, Sichuang
  - Tianjin medical university cancer institute & hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang